CLINICAL TRIAL: NCT00970060
Title: Effectiveness of an Exercise Program on Nerve Function and Cutaneous Nerve Fibers in Adults With Type 2 Diabetes
Brief Title: Exercise and Nerve Function in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patricia Kluding, PhD (Other)
Responsible Party: Sponsor-Investigator, Patricia Kluding, PhD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 11385; GCRC #105 (Other: Clinical and Translational Science Unit)
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Diabetic Neuropathy
Keywords: neuropathy; diabetes
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise program (Experimental): Supervised moderately-intense exercise, including both aerobic and strengthening activities. Sessions are 3-4 days per week for 10 weeks.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Supervised moderately-intense exercise, including both aerobic and strengthening activities. Sessions are 3-4 days per week for 10 weeks.

SUMMARY:
The purpose of this study is to describe the effect of a 10-week exercise program on nerve function and number of nerve fibers in the skin in the lower leg in people with diabetic neuropathy.

DETAILED DESCRIPTION:
The objective for this application is to quantify the benefits of exercise on nerve function including proprioception, and investigate the relationship of these findings with improvements in epidermal and dermal innervation. In this pilot project, we will pursue 2 specific aims: 1) determine the effect of an exercise intervention on nerve function in people with diabetic neuropathy, and 2) assess changes in cutaneous innervation following participation in an exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70
* Type 2 diabetes
* Peripheral neuropathy

Exclusion Criteria:

* Serious cardiac history or other medical problems that would prevent safe participation in exercise

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Quantitative sensory testing | 10 weeks
Nerve conduction studies | 10 weeks
Proprioception | 10 weeks
Dermal and epidermal nerve fiber densities | 10 weeks

SECONDARY OUTCOMES:
Clinical assessments of neuropathy, pain, body mass index, muscle strength, and glycemic control (glycosylated hemoglobin or A1C) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kluding, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Patricia Kluding PhD, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Kluding PM, Pasnoor M, Singh R, Jernigan S, Farmer K, Rucker J, Sharma NK, Wright DE. The effect of exercise on neuropathic symptoms, nerve function, and cutaneous innervation in people with diabetic peripheral neuropathy. J Diabetes Complications. 2012 Sep-Oct;26(5):424-9. doi: 10.1016/j.jdiacomp.2012.05.007. Epub 2012 Jun 18. PMID 22717465